CLINICAL TRIAL: NCT00964691
Title: Intermittent Preventive Treatment With Sulfadoxine-Pyrimethamine Versus Weekly Chloroquine Prophylaxis During Pregnancy in Solomon Islands: a Randomized Controlled Trial
Brief Title: A Randomized Controlled Trial for Intermittent Preventive Treatment in Pregnancy With Fansidar in Solomon Islands
Acronym: IPTpRCT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low prevalence of malaria, high prevalence of reported allergy to sulphur drugs, high proportion of women not meeting the inclusion criterea.
Sponsor: Ministry of Health and Medical Services, Solomon Islands (Other Government)
Collaborators: World Health Organization (Other)
Responsible Party: Dr Lyndes Wini, Ministry of Health and Medical Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01-2009
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Malaria; Malaria in Pregnancy
Keywords: malaria; IPTp; Fansidar; Intermittent Preventive Treatment in pregnancy; pregnancy; prophylaxis; Chloroquine; Anemia; Prevention; Placental malaria; Solomon Islands; Low birth weight
MeSH Terms: conditions — Malaria; Anemia | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chloroquine prophylaxis (Active Comparator): 300 mg weekly by mouth from the enrolment date until delivery. Only the enrolment dose will be supervised.
  Interventions: Drug: Chloroquine prophylaxis
- IPTp with Sulphadoxine-pyrimethamine (Active Comparator): 3 tablets of SP (500 mg sulfadoxine and 25 mg pyrimethamine per tablet) by mouth under supervision at enrolment, and 3 tablets of SP under supervision 4 to 12 weeks later in pregnancy (timing of second dose depends upon gestation at first dose)
  Interventions: Drug: Sulphadoxine-pyrimethamine

INTERVENTIONS:
Drug: Sulphadoxine-pyrimethamine — 3 tablets of SP (500 mg sulfadoxine and 25 mg pyrimethamine per tablet) by mouth under supervision at enrolment, and 3 tablets of SP under supervision 4 to 12 weeks later in pregnancy (timing of second dose depends upon gestation at first dose)
  Other Names: Fansidar; IPTp/SP; SP
  Arms: IPTp with Sulphadoxine-pyrimethamine
Drug: Chloroquine prophylaxis — 300 mg weekly by mouth from the enrolment date until delivery. Only the enrolment dose will be supervised.
  Other Names: CQ
  Arms: Chloroquine prophylaxis

SUMMARY:
The purpose of this study is to assess the effectiveness of intermittent preventive treatment in pregnancy (IPTp) with Sulphadoxine-pyrimethamine compared to chloroquine prophylaxis in Honiara, Solomon Islands for prevention of malaria and it's adverse effects in pregnancy.

DETAILED DESCRIPTION:
Malaria is a major health problem in the Solomon Islands, with an annual estimated incidence of 158 per 1000 population in 2005, and P. falciparum and P. vivax responsible for respectively 71% and 29% of the clinical cases. Not much is known about the burden of malaria in pregnancy and the effectiveness of weekly chloroquine prophylaxis, the national policy for the prevention of malaria in pregnancy. In Honiara, the capital, 42.7% of the pregnant women are anaemic at their first antenatal clinic (ANC) visit. In a national data-base, clinical malaria in pregnancy was associated with an increased risk of anaemia. High levels of chloroquine drug resistance have been reported (67% treatment failure at day 28 in 2001). Among women who attended an ANC in Honiara and had been offered chloroquine prophylaxis, a high low birth weight risk among primigravidae compared to multigravidae was noted. This information indicates that the current policy may not be optimal for the prevention of malaria and its effects in pregnancy. Intermittent preventive treatment (IPTp) with sulfadoxine-pyrimethamine (SP) in pregnancy is an alternative strategy which has been introduced in many malarious countries in sub-Saharan Africa. Studies which compared IPTp with chloroquine prophylaxis in Africa showed that IPTp was more beneficial. Resistance to SP monotherapy in the Solomon islands has not been examined; however, the resistance to the combination of SP and chloroquine is low (< 10%). IPTp with SP has so far not been implemented in a region where P. vivax is common, and the effect of SP on P. vivax is not clear.

We propose a randomized controlled trial to assess the effectiveness of IPTp with SP compared to chloroquine prophylaxis in Honiara, the Solomon Islands. As outcome measures we will examine the effect on anaemia in third trimester, placental malaria, maternal anaemia at the time of delivery, infant birth weight, and prematurity. Outcomes in women allocated IPTp with SP will be compared with those allocated chloroquine prophylaxis. We expect 2504 women from Honiara City Council to participate in the randomised controlled trial. To assess the burden of malaria in pregnancy in other locations women we expect 1000 women to participate in a survey at the time of delivery among women not participating in the trial. At the end of this study, we will know the burden of malaria in pregnancy in Honiara and Guadalcanal, and we will be able to assist in developing evidence based national guidelines for malaria prevention among pregnant women in the Solomon Islands. The information obtained will be important for other areas and countries with a similar epidemiology of malaria in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 15 to 49 years
* Attending ANC clinic for the first time in this pregnancy
* Assigned routine ANC at a HCC health clinic
* Has experienced quickening (feeling the movements of the fetus)
* Gestation of 16 weeks to 32 weeks (as assessed by the last menstrual period [LMP] or by palpation if LMP is not available)
* Willing to adhere to all requirements of study
* Willing to provide informed written consent
* Planning to stay in Honiara for antenatal care and delivery

Exclusion Criteria:

* Used chloroquine prophylaxis in the current pregnancy before this ANC visit
* A history of allergic reaction to sulfa drugs (SP or cotrimoxazole
* Haemoglobin of < 7 g/dl
* Using folic acid in a dose of 5 mg daily (a dose of 1 mg daily or less is acceptable)
* Not willing to adhere to study requirements
* Women who are severely ill

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2504 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Placental malaria among primigravidae at time of delivery | 12 months

SECONDARY OUTCOMES:
Low birth weight among primigravidae | 12 months
Maternal anaemia (Hb <11 g/dl) in the third trimester | 12 months
Maternal anaemia (Hb <11 g/dl) at delivery | 12 months
Malaria parasitemia at delivery | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria van Eijk, MD PhD, Study Chair
Locations (1):
- Honiara City Council, Honiara, Solomon Islands

REFERENCES:
- [Derived] Wini L, Appleyard B, Bobogare A, Pikacha J, Seke J, Tuni M, Hou L, Hii J, McCarthy J, van Eijk AM. Intermittent preventive treatment with sulfadoxine-pyrimethamine versus weekly chloroquine prophylaxis for malaria in pregnancy in Honiara, Solomon Islands: a randomised trial. Malariaworld J. 2013 Jun 29;4:12. doi: 10.5281/zenodo.10894954. eCollection 2013. PMID 38828109